CLINICAL TRIAL: NCT05735275
Title: Safety, Tolerability, Pharmacokinetics, and Efficacy of SHR-A2102, In Subjects With Locally Advanced Or Metastatic Solid Tumor Malignancies: A Phase I Open-Label, One-Arm, Multicenter Study.
Brief Title: A Phase 1 Study of SHR-A2102 in Subjects With Advanced Solid Tumors.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-A2102-I-101
Record Dates: First submitted 2023-01-29; First posted 2023-02-21 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-01

CONDITIONS: Advanced Or Metastatic Solid Tumor Malignancies

STUDY DESIGN:
Intervention Model Description: open, multicenter, Single Group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-A2102 Does Escalation and Expansion (Experimental)
  Interventions: Drug: SHR-A2102

INTERVENTIONS:
Drug: SHR-A2102 — All participants receive SHR-A2102 alone.

SUMMARY:
This is a first in human, open-label, single-arm, multicenter dose escalation and expansion Phase 1 study of SHR-A2102 in patients with advanced or metastatic solid tumors. The purpose of this study is to assess the tolerability, safety, pharmacokinetics and immunogenicity of SHR-A2102 and preliminary anti-tumor efficacy

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and the willingness to sign a written informed consent document；
2. Aged ≥18 years old;
3. Histologically or cytologically confirmed advanced or metastatic malignant tumor;
4. Presence of at least one measurable lesion in agreement to RECIST criteria;
5. Eastern Cooperative Oncology Group (ECOG) performance status 0 to 1;
6. Life expectancy ≥3 months;
7. Adequate organ performance based on laboratory blood tests;
8. Women of childbearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation.

Exclusion Criteria:

1. Previous received anti-cancer systemic therapy including chemo-therapy, radiation therapy, target therapy or immuno-therapy within 4 weeks before the first dose;
2. Previous received experimental medication or therapy within 4 weeks before the first dose;
3. Previous therapeutic surgery within 4 weeks;
4. Has unresolved toxicities from previous anticancer therapy, defined as toxicities not yet resolved to NCI-CTCAE version 5.0 grade ≤ 1.
5. Known allergic to any compound of SHR-A2102;
6. Patients with uncontrolled or active brain metastasis；
7. Patients with clinical significant lung disease;
8. Patients with history of autoimmune diseases;
9. Known active hepatitis B or C infection;
10. Other serious accompanying illnesses, which, in the investigator's assessment, could seriously adversely affect the safety of the treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Estimated)
Dates: Start 2023-03-03 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Dose Limited Toxicity (DLT) | 21 Days (first cycle)
Maximum tolerable dose (MTD) | 21 Days (first cycle)
Recommended dose for phase II (RP2D) | Up to 8 months

SECONDARY OUTCOMES:
Area under the plasma concentration time curve in the dosing interval AUC(TAU) of SHR-A2102 | 30 days after last dose
Maximum observed plasma concentration (Cmax) of SHR-A2102 | 30 days after last dose
Time of maximum observed plasma concentration (Tmax) of SHR-A2102 | 30 days after last dose
Immunogenicity Analysis | 30 days after last dose
  ADA
ORR | 24 months
  Objective Response Rate
DCR | 24 months
  Disease Control Rate
DoR | 24 months
  Duration of Response
PFS | 24 months
  Progression-Free-Survival
OS | 24 months
  Overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided